CLINICAL TRIAL: NCT04311398
Title: Development and Verification of a New Coronavirus Multiplex Nucleic Acid Detection System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Chief of dpartment of infectious disease, Huashan Hospital
Other Study IDs: KY2020-COVID-19
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Respiratory infection group: Patients went to fever clinic with respiratory infectious symptoms in Huashan Hospital affiliated to Fudan University
  Interventions: Diagnostic Test: New QIAstat-Dx fully automatic multiple PCR detection platform

INTERVENTIONS:
Diagnostic Test: New QIAstat-Dx fully automatic multiple PCR detection platform — We use the New QIAstat-Dx fully automatic multiple PCR detection platform to test the enrolled patients

SUMMARY:
Our project intends to independently develop a fully enclosed rapid detection system for a total of 22 pathogens, including SARS-CoV-2, on the basis of the QIAstat-Dx fully automatic multiple PCR detection platform. The reasonably designed experiments are used to verify the performance of the cartridge detection and prove its clinical application value. The 22 pathogens tested in this project includes 4 coronavirus subtypes, A / B flu, parainfluenza virus, respiratory syncytial virus, etc., which is of great significance for the differential diagnosis of similar patients.

DETAILED DESCRIPTION:
COVID-19 has not been well suppressed, and became a pandemic within 3 months globally is mainly because of the virus characteristic in the following aspects:

1. Long incubation period (average 5-7 days, up to 28 days), and the incubation period is contagious
2. Strong transmissibility, virus can be transmitted through aerosol
3. Difficulty distinguishing infected patients from other pathogenic infections
4. High negative rate of nucleic acid detection in upper respiratory tract samples of infected patients, which increases the difficulty of differential diagnosis of infection with other pathogens The existing RT-PCR nucleic acid detection kits for SARS-CoV-2 has two major problems. First, the procedure is not automated leading to higher requirements for personnel operation level and environment sterilize. What's more the kits are SARS-CoV-2 only. Once the test result is negative, it cannot help diagnose the exact pathogen in one time of experiment.

Therefore, this project intends to independently develop a fully enclosed rapid detection system for a total of 22 pathogens, including SARS-CoV-2, on the basis of the QIAstat-Dx fully automatic multiple PCR detection platform. The reasonably designed experiments are used to verify the performance of the cartridge detection and prove its clinical application value. The 22 pathogens tested in this project includes 4 coronavirus subtypes, A / B flu, parainfluenza virus, respiratory syncytial virus, etc., which is of great significance for the differential diagnosis of similar patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients went to the fever clinic with respiratory infectious symptoms

Exclusion Criteria:

* none

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We'd like to enroll the patients who went to the fever clinic with respiratory infectious symptoms in Huashan Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-13 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity， spectivity turnaround time of the New QIAstat-Dx fully automatic multiple PCR detection platform | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No